CLINICAL TRIAL: NCT06459050
Title: Effects of Overcoming Isometric Unilateral Conditioning Activity on Subsequent Single-Leg Drop Jump in Elite and Amateur Volleyball Players
Brief Title: Effects of Isometric Conditioning Activity on Subsequent Jumping Performance in Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Jerzy Kukuczka Academy of Physical Education in Katowice (Other)
Collaborators: Charles University, Czech Republic (Other); University School of Physical Education, Krakow, Poland (Other)
Responsible Party: Principal Investigator, Michal Krzysztofik, PhD, The Jerzy Kukuczka Academy of Physical Education in Katowice
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRIMUS 22/HUM/019
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Resistance Training
Keywords: resistance training; strength and conditioning; physical activity; athletic performance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The study was performed following a randomized, double-blind crossover design, where each participant performed two experimental sessions.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dominant Limb Conditioning Activity (Experimental): Each participant performed a single-leg drop jump for both the dominant and non-dominant limbs before and after completing the CA.
  Interventions: Other: Dominant Limb Overcoming Isometric Conditioning Activity
- Non-dominant Limb Conditioning Activity (Experimental): Each participant performed a single-leg drop jump for both the non-dominant and non-dominant limbs before and after completing the CA.
  Interventions: Other: Non-dominant Limb Overcoming Isometric Conditioning Activity

INTERVENTIONS:
Other: Dominant Limb Overcoming Isometric Conditioning Activity — Each session involved performing 3 sets of 3-second overcoming isometric split squats with a 3-minute rest between sets as a conditioning activity performed by the dominant limb.
  Arms: Dominant Limb Conditioning Activity
Other: Non-dominant Limb Overcoming Isometric Conditioning Activity — Each session involved performing 3 sets of 3-second overcoming isometric split squats with a 3-minute rest between sets as a conditioning activity performed by non-dominant limb.
  Arms: Non-dominant Limb Conditioning Activity

SUMMARY:
The pairing of high-effort exercise, called conditioning activity, with a biomechanically similar high-velocity power movement is considered a valid method to effectively facilitate muscle power adaptations. Research has mainly focused on using this method in exercises performed by both limbs, even though sports tasks are often executed through motion sequences produced by a single limb alternately. However, available studies have focused solely on the dominant leg, leaving it unclear if the effectiveness is similar in both legs and how it transfers between them. Therefore, this study aims to evaluate the immediate effects of the isometric split squat exercise on single-leg drop jump performance in volleyball players, considering their training status.

ELIGIBILITY:
Inclusion Criteria:

* no lower-limb serious injury, including tendon or muscle tear,
* participation in regular resistance training and competition.
* for the elite group participants competed at the highest national volleyball league for at least two consecutive seasons.
* for the amateur group participants competed in junior groups outside the highest league level.

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-02 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Drop Jump Height | Immediately pre- and at 4th and 8th minute post-completion of conditioning activity.
  Drop jump height estimated via take-off velocity performed on force plates. Participants performed 2 trials at each time-point.
Drop Jump Contact Time | Immediately pre- and at 4th and 8th minute post-completion of conditioning activity.
  Drop jump contact time was estimated via time spent on the ground between drop and jump transition performed on force plates. Participants performed 2 trials at each time-point.
Drop Jump Reactive Strength Index | Immediately pre- and at 4th and 8th minute post-completion of conditioning activity.
  Drop jump reactive strength index was estimated via jump height divided by the contact time performed on force plates. Participants performed 2 trials at each time-point.

CONTACTS AND LOCATIONS:
Locations (1):
- The Jerzy Kukuczka Academy of Physcial Education in Katowice, Katowice, Silesian Voivodeship, Poland

REFERENCES:
- [Derived] Terbalyan A, Mikolajec K, Krzysztofik M, Urbanski R, Jarosz J, Stastny P, Spieszny M. Effects of overcoming isometric unilateral conditioning activity on subsequent single-leg drop jump in elite and amateur volleyball players: a randomized crossover trial. BMC Sports Sci Med Rehabil. 2025 Feb 28;17(1):30. doi: 10.1186/s13102-025-01083-9. PMID 40022177